CLINICAL TRIAL: NCT03526315
Title: Antimicrobial Effect of Casein Phosphopeptide Amorphous Calcium Phosphate on Streptococcus Mutans in Children
Brief Title: Antimicrobial Effect of Different Pastes on Streptococcus Mutans in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JUST
Record Dates: First submitted 2017-03-06; First posted 2018-05-16 (Actual); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Mutans Streptococci; Oral Health
Keywords: CPP-ACP paste; Fluoride toothpaste; Combined use of fluoride and CPP-ACP paste; MS reduction; Antibacterial; Children
MeSH Terms: interventions — Fluorides; casein phosphopeptide-amorphous calcium phosphate nanocomplex

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled trial involving 127 children ages between 4 and 5 years. They will be examined and chosen randomly for the study. One hundred and twenty seven children will be divided equally into three groups: Group 1 will use CPP-ACP twice daily, Group 2 will apply fluoride toothpaste twice daily, Group 3 will apply fluoridated toothpaste and CPP-ACP twice daily. Oral swabs will be collected from children to measure MS levels in terms of (CFU) using Saliva Check Mutans kits ( GC, Asia) for this purpose. Samples will be analyzed for MS colonization before antibacterial agent application (baseline) and at 3, and 6 month intervals.
Oversight: Data Monitoring Committee: No

ARMS (3):
- CPP-ACP paste (Active Comparator): Casein phosphopeptide amorphous calcium phosphate is a product that contains calcium, phosphate, protein and casein.
  Interventions: Other: CPP-ACP paste
- Fluoride toothpaste (Active Comparator): Fluoride toothpaste
  Interventions: Other: Fluoride toothpaste
- Both (Fluoride and CPP-ACP) (Active Comparator): Fluoride toothpaste and CPP-ACP paste
  Interventions: Other: Both (Fluoride and CPP-ACP)

INTERVENTIONS:
Other: CPP-ACP paste — Children will brush their teeth with CPP-ACP paste twice daily.
  Arms: CPP-ACP paste
Other: Fluoride toothpaste — Children will brush their teeth with fluoridated toothpaste twice daily.
  Arms: Fluoride toothpaste
Other: Both (Fluoride and CPP-ACP) — Children will brush their teeth with fluoridated toothpaste and apply CPP-ACP immediately after tooth brushing, twice daily.
  Arms: Both (Fluoride and CPP-ACP)

SUMMARY:
This study is a randomized controlled trial involving 127 children ages between 4 and 5 years to investigate the efficacy of Casein Phosphopeptide-Amorphous Calcium Phosphate (CPP-ACP) in reducing Streptococcus mutans (S. mutans) bacteria, and compare that with fluoride alone, or combined use of fluoride and CPP-ACP over a 6 month period using Saliva Check Mutans kits to detect Mutans Streptococci (MS). It is expected that all used anti-cariogenic agents will have the ability to reduce the S. mutans level in different values.

DETAILED DESCRIPTION:
Aim: The aim of this study is to investigate the efficacy of CPP-ACP in reducing S. mutans, and compare that with fluoride alone, or combined use of fluoride and CPP-ACP.

Materials and methods: This study is a randomized controlled trial involving 127 children ages between 4 and 5 years. They will be examined and chosen randomly for the study. One hundred and twenty seven children will be divided equally into three groups: Group 1 will use CPP-ACP twice daily, Group 2 will apply fluoride toothpaste twice daily, Group 3 will apply fluoridated toothpaste and CPP-ACP twice daily. Oral swabs will be collected from children to measure S. mutans levels in terms of Colony forming units (CFU) using Saliva Check Mutans kits (GC© , Asia) for this purpose. Samples will be analyzed for S. mutans colonization before antibacterial agent application (baseline) and at 3, and 6 month intervals.

Expected results: it is expected that all used anti-cariogenic agents will have the ability to reduce the S. mutans levels in different levels.

ELIGIBILITY:
Inclusion Criteria:

* Healthy 4-5 years old children, with primary dentition, and early childhood caries/high risk caries

Exclusion Criteria:

* Milk protein (casein) sensitivity
* Patient who has taken antibiotics in the last month
* Lack in cooperation in oral examination
* Medically compromised children
* Children that have received fluoride supplement or professional topical fluoride application at least three months before or during the study period.

Ages: 4 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 127 (Actual)
Dates: Start 2016-03; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Changes in Streptococcus mutans levels (Colony Forming Units/CFU) using Saliva Check Mutans kits ( GC, Asia) | 3 and 6 months
  Changes in Streptococcus mutans after use of CPP-ACP, Fluoride or both Saliva Check Mutans kits ( GC, Asia)

SECONDARY OUTCOMES:
Changes in caries using the decayed, missing due to caries, filled, deciduous teeth (dmft index) | 3 and 6 months
  Changes in dmft after use of CPP-ACP, Fluoride or both agents over 3 and 6 months.
Changes in caries using the decayed, missing due to caries, filled, deciduous tooth surfaces (dmfs) index | 3 and 6 months
  Changes in dmfs after use of CPP-ACP, Fluoride or both agents over 3 and 6 months.
Changes in caries using the International Caries Detection and Assessment System (ICDAS) scores | 3 and 6 months
  Changes in ICDAS scores over 3 and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Ola Al-Batayneh, MDSc, FRACDS, Principal Investigator — Associate Professor in Pediatric Dentistry
Locations (1):
- Jordan University of Science and Technology, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No
The data will be shared as in demographics of the study sample.